CLINICAL TRIAL: NCT04569396
Title: Effect of Bariatric Surgery on Fatty Liver Disease. A Prospective One-Year Follow-Up Study
Brief Title: Bariatric Surgery and Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: CHIR-06-Fatty_Liver; SGS03/LF/2018 (Other Grant/Funding Number: University of Ostrava)
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Morbid Obesity; Diabetes; Hypertension
Keywords: non-alcoholic fatty liver disease; bariatric surgery; obesity; liver fibrosis
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus; Hypertension; Non-alcoholic Fatty Liver Disease; Obesity; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Alcoholic Fatty Liver Disease: A total of 72 severely or morbidly obese patients with non-alcoholic fatty liver disease and associated co-morbidities like diabetes and hypertension were enrolled into the study.
  Interventions: Diagnostic Test: Biochemistry analysis; Diagnostic Test: NAFLD fibrosis score; Other: BMI measurement; Diagnostic Test: Fibrosis 4 Index; Diagnostic Test: Fatty Liver Index

INTERVENTIONS:
Diagnostic Test: Biochemistry analysis — Biochemistry analysis of liver parameters were analyzed among the study subjects before and after the surgery.
Diagnostic Test: NAFLD fibrosis score — NAFLD fibrosis score was determined among the study subjects before and after the surgery.
Other: BMI measurement — BMI was measured among the study subjects before and after the surgery.
Diagnostic Test: Fibrosis 4 Index — Fibrosis 4 Index was determined among the study subjects before and after the surgery.
Diagnostic Test: Fatty Liver Index — Fatty Liver Index was determined among the study subjects before and after the surgery.

SUMMARY:
The study is based on data from morbidly obese patients who fulfilled the criteria for bariatric surgery during 2016-2018 at the Department of Surgery, University Hospital Ostrava, Czech Republic.

DETAILED DESCRIPTION:
The study is based on data from morbidly obese patients who fulfilled the criteria for bariatric surgery during 2016-2018 at the Department of Surgery, University Hospital Ostrava, Czech Republic. Patients with age above 18 years, BMI > 35-40 kg/m2, and associated with at least one of the complications including hypertension, diabetes, and failure of the current therapies to relieve the symptoms were included in the study. Patients included in the current study do not have a history of excessive alcohol consumption, use of hepatotoxic drugs, infectious liver diseases (i.e. hepatitis A, B, C), and genetic hemochromatosis. A total of 72 patients including n = 26 during 2016, n = 26 during 2017, and n = 20 during 2018 who qualified for bariatric surgeries were included in this observational study. Data related to patients' gender, age (years), weight (kg), height (cm), and associated co-morbidities like diabetes and hypertension were recorded before surgery. BMI (kg/m2), biochemical parameters including triglycerides profile (mmol/L), platelet count (number/L), Gamma glutamyl-transferase (international units - IU/L), albumin concentration (g/L), Alanine amino-transferases (units/L), Aspartate aminotransferases (international units - IU/L), were evaluated following standard procedures. Platelet count, triglycerides, and enzymes were determined using standard procedures.

The biochemical results were compared to the corresponding paired values before surgery and after surgery. The current study was designed to prospectively investigate the effect of bariatric surgeries among non-alcoholic obese individuals from 2016-2018 and one year follow up on liver biochemistry, BMI, non-alcoholic fatty liver disease (NAFLD) fibrosis score, Fibrosis 4 (FIB 4) Index, and Fatty Liver Index (FLI).

The continuous variables were expressed as mean ± standard deviation and median (interquartile range) in case of normal and non-normal distribution, respectively. The Shapiro-Wilk test was used to test for normal distribution. The within-patient changes in clinical parameters (continuous or ordinal variables) from baseline to 1-year after bariatric surgery were compared using the Wilcoxon matched-pairs signed-rank tests for ordinal variables and continuous variables when the change was not normal or using the paired Student's t-test otherwise. The statistical testing was done at the two-tailed α level of 0.05. The data were analyzed using GraphPad Prism Version 8.0.2 (GraphPad Software, Inc., USA).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and above
* BMI > 35-40 kg/m2
* hypertension or diabetes or failure of the current therapies to relive the symptoms

Exclusion Criteria:

* history of excessive alcohol consumption
* use of hepatotoxic drugs
* infectious liver diseases (i.e. hepatitis A, B, C)
* genetic hemochromatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age above 18 years, BMI > 35-40 kg/m2 and associated with at least one of the complications including hypertension, diabetes and failure of the current therapies to relive the symptoms were included in the study. Patients included in the current study does not have a history of excessive alcohol consumption, use of hepatotoxic drugs, infectious liver diseases (i.e. hepatitis A, B, C) and genetic hemochromatosis.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2018-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Biochemistry analysis | 1 year
  Biochemistry analysis of liver parameters were analyzed among the study subjects before and after the surgery (for details please see the Detailed description of the study)
Non-Alcoholic Fatty Liver Disease (NAFLD) fibrosis score | 1 year
  NAFLD fibrosis score was determined among the study subjects before and after the surgery.
BMI measurement | 1 year
  BMI was measured among the study subjects before and after the surgery.
Fibrosis 4 Index | 1 year
  Fibrosis 4 Index was determined among the study subjects before and after the surgery.
Fatty Liver Index | 1 year
  Fatty Liver Index was determined among the study subjects before and after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Toman, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be made available to other researchers upon request.

REFERENCES:
- [Derived] Toman D, Vavra P, Jelinek P, Ostruszka P, Ihnat P, Foltys A, Pelikan A, Roman J. Effect of bariatric surgery on fatty liver disease in obese patients: A prospective one year follow-up study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2022 May;166(2):195-203. doi: 10.5507/bp.2021.021. Epub 2021 Apr 19. PMID 33885048